CLINICAL TRIAL: NCT02867345
Title: A Dose-escalation Phase I Trial of PD-1 Knockout Engineered T Cells for the Treatment of Castration Resistant Prostate Cancer
Brief Title: PD-1 Knockout Engineered T Cells for Castration Resistant Prostate Cancer
Status: Withdrawn | Type: Observational
Why Stopped: no funding or finacial support
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Wujiang Liu, Professor, Peking University
Other Study IDs: 11007965939
Record Dates: First submitted 2016-08-11; First posted 2016-08-15 (Estimated); Last update posted 2019-03-06 (Actual); Status verified 2016-08

CONDITIONS: Hormone Refractory Prostate Cancer
MeSH Terms: interventions — Cyclophosphamide; Interleukin-2

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Test group: Peripheral blood lymphocytes will be collected and Programmed cell death protein 1(PDCD1) gene will be knocked out by CRISPR Cas9 in the laboratory (PD-1 Knockout T cells). The lymphocytes will be selected and expanded ex vivo and infused back into patients. Cyclophosphamide at 20mg/kg single dose will be administered 3 days i.v. before cell infusion. A total of 2 x 10^7/kg PD-1 Knockout T cells will be infused in one cycle. Each cycle is divided into three administrations, with 20% infused in the first administration, 30% in the second, and the remaining 50% in the third.Interleukin-2 (IL-2) will be given in the following 5 days, 720000 international unit（IU）/Kg/ day (if tolerant). Patients will receive a total of 2, 3, 4 cycles of treatment.
  Interventions: Biological: PD-1 Knockout T Cells; Drug: Cyclophosphamide; Drug: IL-2
- Comparable group: Peripheral blood lymphocytes will be collected and Programmed cell death protein 1(PDCD1) gene will not be knocked out by CRISPR Cas9 in the laboratory (PD-1 Wild-type T cells). The lymphocytes will be selected and expanded ex vivo and infused back into patients. Cyclophosphamide at 20mg/kg single dose will be administered 3 days i.v. before cell infusion. A total of 2 x 10^7/kg PD-1 wild-type T cells will be infused in one cycle. Each cycle is divided into three administrations, with 20% infused in the first administration, 30% in the second, and the remaining 50% in the third. Interleukin-2 (IL-2) will be given in the following 5 days, 720000 international unit（IU）/Kg/day (if tolerant).
  Interventions: Drug: Cyclophosphamide; Drug: IL-2

INTERVENTIONS:
Biological: PD-1 Knockout T Cells — PD-1 Knockout T Cells and PD-1 wild-type T Cells will be made by Cell Biotech Co., Ltd. 2x107/kg T cells will be used for test group and comparable group separately.
  Groups: Test group
Drug: Cyclophosphamide — Cyclophosphamide at 20mg/kg single dose will be administered 3 days i.v. before cell infusion.
  Interleukin-2 (IL-2) will be given in the following 5 days, 720000 international unit（IU）/Kg/day (if tolerant).
  Other Names: cytophosphane
Drug: IL-2 — Interleukin-2 (IL-2) will be given in the following 5 days after cell infusion, 720000 international unit（IU）/Kg/ day (if tolerant).
  Other Names: Interleukin-2 (IL-2)

SUMMARY:
This study will evaluate the safety of PD-1 knockout engineered T cells in treating castration resistant prostate cancer (CRPC). Blood samples will also be collected for research purposes.

DETAILED DESCRIPTION:
This is a dose-escalation study of ex-vivo knocked-out, expanded, and selected PD-1 knockout-T cells from autologous origin. Patients are assigned to 1 of 3 treatment groups to determine the maximal tolerant dose. After the lower number of cycles are considered tolerant, an arm of the next higher number of cycles will be open to next patients. Biomarkers and immunological markers are collected and analyzed as well.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically and clinical verified castration resistant prostate cancer with measurable lesions (On CT: longest diameter of tumoral lesion >=10 mm, shorted diameter of lymph node >=15 mm; measurable lesions should not have been irradiated)
* Progressed after all standard treatment
* Performance score: 0-1
* Expected life span: >= 6 months
* Toxicities from prior treatment has resolved. Washout period is 4 weeks for chemotherapy, and 2 weeks for targeted therapy
* Major organs function normally
* Willing and able to provide informed consent

Exclusion Criteria:

* Pathology is mixed type
* Emergent treatment of tumor emergency is needed
* Poor vasculature
* Coagulopathy, or ongoing thrombolytics and/or anticoagulation
* Blood-borne infectious disease, e.g. hepatitis B
* History of mandatory custody because of psychosis or other psychological disease inappropriate for treatment deemed by treating physician
* With other immune diseases, or chronic use of immunosuppressants or steroids
* Compliance cannot be expected
* Other conditions requiring exclusion deemed by physician

Ages: 45 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-11; Primary Completion 2020-11 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants with Adverse Events and/or Dose Limiting Toxicities as a Measure of Safety and tolerability of dose of PD-1 Knockout T cells using Common Terminology Criteria for Adverse Events (CTCAE v4.0) in patients | Dose Escalation - Approximately 6 months

SECONDARY OUTCOMES:
Response Rate:Response will be evaluated according to RECIST v1.1 | 90 days
Progression free survival - PFS | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to average 10 months
Overall Survival - OS | The time from randomization to death from any cause, assessed up to 2 years
Peripheral blood circulating tumor DNA | 6 weeks
Temporal Interleukin-2 change in the peripheral blood | Baseline and 1 month and 3 months
Temporal Interferon-γ change in the peripheral blood | Baseline and 1 month and 3 months
Temporal Interleukin-6 change in the peripheral blood | Baseline and 1 month and 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Urology Peking University First Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided
Plan to open

REFERENCES:
- [Background] Taube JM. Unleashing the immune system: PD-1 and PD-Ls in the pre-treatment tumor microenvironment and correlation with response to PD-1/PD-L1 blockade. Oncoimmunology. 2014 Dec 21;3(11):e963413. doi: 10.4161/21624011.2014.963413. eCollection 2014 Nov. PMID 25914862
- [Background] Yatsuda J, Eto M. [Current status and prospects of immunotherapy for castration-resistant prostate cancer]. Nihon Rinsho. 2014 Dec;72(12):2174-8. Japanese. PMID 25518354
- [Result] Modena A, Ciccarese C, Iacovelli R, Brunelli M, Montironi R, Fiorentino M, Tortora G, Massari F. Immune Checkpoint Inhibitors and Prostate Cancer: A New Frontier? Oncol Rev. 2016 Apr 15;10(1):293. doi: 10.4081/oncol.2016.293. eCollection 2016 Apr 15. PMID 27471580
- [Result] Bishop JL, Sio A, Angeles A, Roberts ME, Azad AA, Chi KN, Zoubeidi A. PD-L1 is highly expressed in Enzalutamide resistant prostate cancer. Oncotarget. 2015 Jan 1;6(1):234-42. doi: 10.18632/oncotarget.2703. PMID 25428917
- [Derived] Yi L, Li J. CRISPR-Cas9 therapeutics in cancer: promising strategies and present challenges. Biochim Biophys Acta. 2016 Dec;1866(2):197-207. doi: 10.1016/j.bbcan.2016.09.002. Epub 2016 Sep 15. PMID 27641687